CLINICAL TRIAL: NCT02721030
Title: Mbarara Acute Heart Failure Registry: Opportunities to Improve Care of Patients Hospitalized With Acute Decompensated Heart Failure in Mbarara Regional Referral Hospital, Uganda
Brief Title: Mbarara Acute Heart Failure Registry
Acronym: MAHFER
Status: Completed | Type: Observational
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Virginia (Other); Abbott Point of Care (Industry)
Responsible Party: Principal Investigator, Samson Okello, Clinical Lecturer/Epidemiologist, Mbarara University of Science and Technology
Other Study IDs: 26/11-14
Record Dates: First submitted 2016-03-16; First posted 2016-03-28 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Heartfailure
Keywords: Heartfailure; 1-year mortality; heartfailure quality of life; sub-Saharan Africa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective cohort to describe clinical characteristics, predictors of poor outcomes both during hospitalization and at home, functional status, and quality of life among patients aged 13 years or more, consecutively admitted with acute decompensated heart failure at Mbarara Regional Referral Hospital.

DETAILED DESCRIPTION:
This is a prospective observational cohort study to collect comprehensive data of heartfailure patients during and after hospitalization for acute heart failure at Mbarara Regional Referral Hospital (MRRH), Uganda. The investigators will collect sociodemographic, clinical, quality of life, functional status, and clinical cardiovascular disease measures during hospitalization and follow up for up to 1 year from the date of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with a confirmed clinical diagnosis of acute heartfailure aged 13 years or above at Mbarara Regional Referral Hospital, Uganda

Exclusion Criteria:

* Body swelling from kidney disease, liver disease or malnutrition.
* Acute kidney disease with no previous history/documentation of heart disease.
* History suggestive of chronic kidney disease with no previous history/documentation of heart disease.
* History suggestive of chronic liver disease with no previous history/documentation of heart disease.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target Population: Patients hospitalized in a medical ward of a resource poor setting.
  Accessible Population: Patients aged 13 years or more admitted with a diagnosis of acute decompensated Heart failure to the Medical ward of Mbarara Regional Referral Hospital.
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 1 year

SECONDARY OUTCOMES:
Length of hospitalization | 1 year
  Length of hospital stay
Quality of life using the SF-36 questionnaire | 1 year
  Quality of life will be measured using SF-36 questionnaire.
Functional status using the Kansas city cardiomyopathy questionnaire | 1 year
  Kansas city cardiomyopathy questionnaire will be used to measure functional status during hospitalization and quarterly after hospitalization with acute heartfailure.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Fardous, MMED, Study Director — Mbarara University of Science & Technology
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, N/A = Not Applicable, Uganda

IPD SHARING:
Plan to Share IPD: No
Not indicated

REFERENCES:
- [Result] Abeya FC, Lumori BAE, Akello SJ, Annex BH, Buda AJ, Okello S. Incidence and predictors of 6 months mortality after an acute heart failure event in rural Uganda: The Mbarara Heart Failure Registry (MAHFER). Int J Cardiol. 2018 Aug 1;264:113-117. doi: 10.1016/j.ijcard.2018.03.110. Epub 2018 Mar 29. PMID 29655949